CLINICAL TRIAL: NCT06649825
Title: Evaluation of the Efficacy of Vitamin B1 in Patients with Familial Adenomatous Polyposis: an Exploratory Study
Brief Title: Efficacy of Vitamin B1 in Familial Adenomatous Polyposis Patients.
Acronym: VitB1; FAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiZhongshanEndoscopy2
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Familial Adenomatous Polyposis (FAP)
Keywords: Familial adenomatous polyposis; thiamin
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin B1 (Experimental)
  Interventions: Drug: Vitamin B1

INTERVENTIONS:
Drug: Vitamin B1 — Vitamin B1 tablets, 100mg bid, taken orally for one year

SUMMARY:
This study aimed to investigate the efficacy of vitamin B1 in patients with familial adenomatous polyposis, and to determine the inhibitory effect of vitamin B1 on the size and number of colorectal adenomas by administering oral vitamin B1 therapy for 1 year and colonoscopy follow-up every 3 months

DETAILED DESCRIPTION:
We will mark a region with a diameter of no more than 5 cm, containing at least 3 polyps, each with a diameter of 5-15 mm. Continuous video recording will be conducted throughout the colonoscopy procedure to provide baseline reference images of the colorectal polyps. Patients with familial adenomatous polyposis were given 100mg bid dose of vitamin B1 orally for one year, and colonoscopies were followed every 3 months to observe changes in the size and number of polyps in the designated area.

ELIGIBILITY:
Inclusion Criteria

1. Patients with a confirmed diagnosis of classical familial adenomatous polyposis (FAP) based on colonoscopy, histopathology, and genetic testing.
2. Aged between 18 and 80 years, with no restriction on gender.
3. No history of total colectomy, with remaining bowel segments available for evaluation.
4. Presence of more than 10 adenomatous polyps in the colon or rectum.
5. Normal liver and kidney function.
6. Willing to participate in vitamin B1 therapy and commit to regular follow-up appointments.

Exclusion Criteria

1. Use of medications for more than one week in the past three months, or inability to avoid continuous use during the study period, that may affect colorectal polyps, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), ω-3 polyunsaturated fatty acids, rapamycin, and curcumin.
2. Use of medications for more than one week in the past three months, or inability to avoid continuous use during the study period, that may affect vitamin B1 absorption, metabolism, or excretion, including aminoglycoside antibiotics, thiazide diuretics, oral contraceptives, antiepileptic drugs, and antituberculosis drugs.
3. Attenuated familial adenomatous polyposis (AFAP).
4. Allergy to vitamin B1.
5. Contraindications to vitamin B1, such as liver or kidney dysfunction, or severe neuropsychiatric disorders.
6. History of total colectomy, with no remaining bowel segments.
7. Pregnant or breastfeeding individuals.
8. Presence of advanced colorectal cancer or metastatic cancer in other locations.
9. Previous radiotherapy, chemotherapy, or tumor immunotherapy.
10. History of alcohol or other substance abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sum of polyp diameters in the delineated area | 3 months
  The diameter of each polyp was assessed by two independent endoscopists and the average of two diameters perpendicular to each other was reported. The diameter of the polyp was determined with reference to the titanium clip, blood vessels and scar in the visual field.

SECONDARY OUTCOMES:
The number of polyps in the delineated area | 3 months
  The number of polyps was assessed by two independent endoscopists, and disputes were decided by a third endoscopist
Levels of vitamin B1-associated metabolites, including TMP, TPP, TTP, and free thiamine, in blood and urine samples and in polyps outside the delineated area | 3 months
  The content of vitamin B1 related metabolites was determined by liquid chromatography-tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Pinghong Zhou, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Original data could be shared at request by email after publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be available after publication of the study
Access Criteria: The shared data could be available by contacting Dr. Xin-Yang Liu at liu.xinyang@zs-hospital.sh.cn.